CLINICAL TRIAL: NCT07018895
Title: Safety and Efficacy of Intermittent hypoxiс-hyperoxiс Personalized Training Sessions for the Creation of an Organoprotective Phenotype in Elderly People SHIELD
Brief Title: Personalized Hypoxic-hyperoxic Preconditioning in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Nikolay Kamenshchikov, Principal Investigator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SHIELD
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Preconditioning
Keywords: OXYTERRA; intermittent hypoxic-hyperoxic training; cerebral tissue oxygenation
MeSH Terms: interventions — Particulate Matter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): ambient air (FiO2 = 21%) will be delivered for 3 days 1 time a day for 45 minutes
  Interventions: Drug: Sham treatment
- Main group (Experimental): FiO2 reduced by 20% will be delivered for 6 minutes alternating with 34% FiO2 for 3 minutes (45 minutes in total as 5 full circles) within 3 days 1 time a day
  Interventions: Drug: FiO2 reduced by 20% alternating with 34% FiO2

INTERVENTIONS:
Drug: Sham treatment — ambient air (FiO2 = 21%) will be delivered for 3 days 1 time a day for 45 minutes
  Other Names: ambient air
  Arms: Control group
Drug: FiO2 reduced by 20% alternating with 34% FiO2 — FiO2 reduced by 20% alternating with 34% FiO2
  Other Names: FiO2
  Arms: Main group

SUMMARY:
This study investigates an original protocol of personalized hypoxic-hyperoxic preconditioning utilizing a personalized approach on the basis of cerebral tissue oxygenation assessed with near-infrared spectroscopy. 20 healthy elderly volunteers will be randomized into two equal groups. Subjects of the experimental group will undergo personalized sessions of intermittent hypoxic-hyperoxic training (IHHT) based on the cerebral tissue oximetry index assessed with near-infrared spectroscopy with a target reduction of 20%. Subjects of the control group (sham treatment) will undergo placebo procedures with atmospheric air.

DETAILED DESCRIPTION:
1. Rationale for the study conduction Chronic diseases, surgical interventions, aging and the effects of drugs and environmental factors have an adverse health effect on the human body. Therefore, the development of novel techniques and improvement of existing methods for organ protection and health preservation is one of the most crucial tasks of modern medicine.

   The term preconditioning refers to describing the phenomenon of increasing the tolerance of a cell, tissue, organ or organism as a whole to the effects of a damaging factor (e.g., ischemia, hypoxia, surgical trauma) as a result of preliminary exposure to sub-damaging stress stimuli. There are various approaches to the implementation of this phenomenon including ischemic preconditioning, pharmacological preconditioning, hypoxic preconditioning and remote preconditioning.

   Of great interest is the concept of hypoxic preconditioning in which the body is deprived of adequate oxygen supply at the tissue level, which contributes to the implementation of a protective phenotype in all organs and tissues. In practice, this technique is usually implemented as an intermittent delivery of hypoxic and normoxic gas mixtures, but recently its modification in which the normoxic phase is replaced by a hyperoxic one has become popular. The method demonstrates promising results, but is not applicable in practice, since most of the completed studies analyze IHHT sessions as a long-term therapy, which is not feasible in a hospital setting.

   The major task is selecting the optimal mode demonstrating both efficacy and feasibility as well as personalizing the IHHT, which justifies the need for this study.
2. Known and potential risks for the study Subjects This is a prospective, single-blind, randomized, placebo-controlled study. This study will include subjects without serious chronic diseases or with diseases during the compensatory stage; therefore the therapy does not carry potential risks. This is confirmed by Uzun et al., 2023, whose systematic review assessed the outcomes of 16 studies of IHHT and intermittent hypoxic-normoxic training conducted on patients with various diseases.

   Since the sessions will be personalized according to cerebral tissue oximetry utilizing near-infrared spectroscopy with a target reduction of 20% in the hypoxic phase of the session, such adverse reactions as impaired consciousness up to the onset of a syncope are possible, as this variable has not been previously assessed in IHHT.

   Due to the absence of serious pathologies in potential study subjects, the potential benefit will be of a general health-improving nature (increased performance, accelerated metabolism and enhanced nervous system).
3. The route of drug administration, dosage, dosing regimen and course of treatment

The dosing regimen for using IHHT should be personalized in each specific case and meet the following criteria:

1. Safety/tolerability for the procedure. 2. Efficacy. 3. Applicability in real clinical practice.

4. Conducting sessions of intermittent hypoxic-hyperoxic training and sham treatment.

The IHHT sessions will utilize the OXYTERRA PRO device (OOO Oxyterra, Russia). This machine generates a gas mixture with 7-16% FiO2 (fraction of inspired oxygen) in the hypoxia phase and 25-33% FiO2 in the hyperoxia phase. The device monitors respiratory rate and respiratory minute volume. The maximum flow rate of the delivered gas mixture is 25 L/min. The IHHT session duration is up to 120 minutes. The device is equipped with a pulse oximeter. In addition, a capnograph will be built into the breathing circuit.

The IHHT sessions will be conducted for 3 days. Before the first IHHT session, each subject will undergo a hypoxic test, which is crucial to identify the required FiO2 level for reducing cerebral tissue oxygenation based on near-infrared spectroscopy by 20% from the baseline.

Conducting a hypoxic test.

1. placing the subject in a supine position;
2. adjusting monitoring of electrocardiogram, SpO2, cerebral oximetry and blood pressure;
3. filling the breathing circuit with a normoxic mixture, connecting the patient to the circuit through an oronasal mask and then fixing it;
4. stepwise reduction in FiO2 (starting from 12% with a step of 0.5% lasting 3 min) until cerebral tissue oxygenation based on near-infrared spectroscopy decreases by 20% from the baseline;
5. FiO2 recording;
6. hyperoxia for 2 min;
7. hypoxic test is completed. Subjects of the control group will receive inhalations of atmospheric air for 6 minutes through the OXYTERRA PRO device instead of a hypoxic test.

IHHT sessions will be carried as follows:

1) placing the subject in a supine position or right/left lateral recumbent; 2) adjusting monitoring of electrocardiogram, SpO2, cerebral oximetry, blood pressure and BIS; 3) filling the breathing circuit with a normoxic gas mixture, connecting the patient to the circuit through an oronasal mask and then fixing it; 4) reduction in FiO2 to the value required for reducing cerebral tissue oxygenation based on near-infrared spectroscopy by 20% from the baseline; 5) hypoxia for 6 min; 6) initiation of hyperoxia with 34% FiO2 for 3 minutes; 7) alternation of hypoxic and hyperoxic phases of the session for 45 minutes (5 full cycles of hypoxic-hyperoxic training).

If necessary, during each hypoxic phase FiO2 will be adjusted to ensure a decrease in cerebral tissue oxygenation based on near-infrared spectroscopy by 20% from the baseline.

During each procedure, study participants will be scrupulously interviewed to identify any adverse effects of the procedure.

Criteria for discontinuation and further termination of IHHT sessions:

1. Individual intolerance to IHHT sessions (discomfort that does not allow the Subject to continue the IHHT sessions).

2. Development of any complications of IHHT sessions:

1. disorder of consciousness;
2. the state of syncope;
3. development of any other life-threatening condition. Sham treatment (placebo procedures) will be performed similarly to IHHT sessions, however, during the entire placebo procedure, ambient air (FiO2 = 21%) will be delivered to the Subjects.

Subjects' participation in the study is supposed to last 4 days. Day 1: clinical and demographic data collection, general medical examination, eligibility criteria assessment, signing of informed consent, randomization, pre-procedural venous blood sampling, ultrasound examination of cerebral hemodynamics, hypoxic test (or inhalation of atmospheric air for patients in the control group), IHHT session #1 (or placebo procedure), observation for one hour.

Day 2: collecting data on the Subject condition for the last 24 hours, IHHT session #2 (or placebo procedure), observation for one hour.

Day 3: collecting data on the Subject condition for the last 24 hours, IHHT session #3 (or placebo procedure), collecting venous blood after the session, observation for one hour.

Day 4: collecting data on the Subject condition for the last 24 hours, ultrasound of cerebral hemodynamics, collecting venous blood.

5. Premature discontinuation of the parts of the study, or termination the study as a whole

The criteria for individual discontinuation of the study and subsequent termination of IHHT sessions will be as follows:

1. Failure in reducing cerebral tissue oxygenation by 20% from the baseline during the hypoxic test.
2. Individual intolerance to IHHT sessions.
3. Development of any complications of IHHT sessions:

1) disorder of consciousness; 2) the state of syncope; 3) development of any other life-threatening condition. The study will be discontinued prematurely if 2 study subjects meet criteria 2 and/or 3 for individual premature discontinuation and are withdrawn from the study.

6. Randomization The subjects will be allocated to 2 equal groups (n=10 in each group). The randomization sequence will be generated in advance using the block randomization (https://www.sealedenvelope.com/) by an independent researcher who will not be involved in conducting IHHT sessions and placebo procedures. Randomization codes (which will match the subjects' belonging to the study groups) will be sealed in sequentially numbered opaque envelopes. The sequential numbers of the envelopes will serve as randomization numbers, which will be recorded in the case report form (CRF) and used if necessary, for instance, in the treatment of complications.

7. Blinding Subjects, investigators, and other staff involved in the interpretation of the results will be blinded to the nature of the intervention until the study is completed. The investigator responsible for conducting IHHT and placebo sessions will remain unblinded and will open the envelope containing information about the subject's study group assignment, and will be responsible for equipment masking, monitoring, and safety of the procedures. IHHT and placebo sessions will be conducted using the same equipment.

8. Ethics General Principles for Protecting the Rights and Health of Research Subjects This study will be conducted in accordance with current regulations and guidelines for clinical trials, including the World Medical Association Declaration of Helsinki, the international standard ICH E6 "Good Clinical Practice," Federal Law No. 323-FZ of November 21, 2011, "On the Fundamentals of Health Protection of Citizens in the Russian Federation," Order of the Ministry of Health of the Russian Federation No. 200n of April 1, 2016, "On the Approval of the Rules of Good Clinical Practice." Before the start of the clinical study, information on this study, including the study protocol, the patient informed consent form, information on the researchers' experience in relevant specialties and their experience in conducting clinical trials, will be submitted to the Biomedical Ethics Committee of Cardiology Research Institute of the Tomsk National Research Medical Center (Tomsk NRMC) for ethical review. The study will begin only after obtaining approval from the Biomedical Ethics Committee, which will also monitor compliance with ethical standards during the conduct of this study and the rights of study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-74 years.
2. Signed informed consent.

Non-inclusion criteria

1. Charlson Comorbidity Index ≤ 3 (with a score of 1 or more on all criteria except for the age factor).
2. Conditions associated with chronic hypoxia or hyperoxia.
3. Uncompensated coronary artery disease.
4. Chronic diseases in the acute or decompensated phase.

Exclusion Criteria:

1. Withdrawal from further participation in the study (revocation of informed consent), unrelated to any of the subsequent points.
2. Inability to reduce cerebral tissue saturation by 20% from baseline during the hypoxic test.
3. Individual intolerance to IHHT sessions.
4. Development of one of the following complications during IHHT sessions:

1). Disorder of consciousness. 2). The state of syncope. 3). Development of any other life-threatening condition.

The fact and the reason for the Subject to be excluded from the study will be recorded in the CRF (Case Report Form), along with all data collected during the study, for further analysis, if planned.

If exclusion occurs according to points 1 and 2 of the exclusion criteria, the subject will be replaced with another participant. If exclusion occurs according to any of the subsequent points, replacement will not be performed.

If exclusion occurs according to points 3 and 4, patients will be thoroughly examined and remain under the observation of the study physicians until their condition is stabilized

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Incidence of intolerance to IHHT sessions (a combined endpoint including individual intolerance showing discomfort that does not allow the Subject to continue the IHHT sessions and/or the incidence of one of the complications of IHHT sessions (disorde | Periprocedural
  The difference in the incidence of intolerance to IHHT sessions (percent)

SECONDARY OUTCOMES:
Systolic blood pressure levels (SBP) (mmHg) | 6, 9, 15, 18, 24, 27, 33, 36, and 45 minutes from the initiation of the IHHT session
  The difference in the levels of SBP during IHHT sessions
Diastolic blood pressure levels (DBP) (mmHg). | 6, 9, 15, 18, 24, 27, 33, 36, and 45 minutes from the initiation of the IHHT session
  The difference in the levels of DBP during IHHT sessions
Heart rate (HR) (bpm) | 6, 9, 15, 18, 24, 27, 33, 36, and 45 minutes from the initiation of the IHHT session
  The difference in HR is assessed in beats per minute
Saturation of peripheral oxygen (SpO2) levels (percentage) | 6, 9, 15, 18, 24, 27, 33, 36, and 45 minutes from the initiation of the IHHT session
  The difference in the levels of SpO2 during IHHT sessions
Respiratory rate (RR) (brpm) | 6, 9, 15, 18, 24, 27, 33, 36, and 45 minutes from the initiation of the IHHT session
  The difference in RR is assessed in breaths per minute The difference in respiratory rate during IHHT sessions
End tidal carbon dioxide (etCO2) levels (mmHg) | 6, 9, 15, 18, 24, 27, 33, 36, and 45 minutes from the initiation of the IHHT session
  The difference in the levels of etCO2 during IHHT sessions The difference in the levels of etCO2 is assessed in mmHg
Incidence of intolerance to IHHT sessions (percent) | Periprocedural
  The difference in the incidence of intolerance to IHHT sessions
Incidence of one of the complications of IHHT sessions (percent) | Periprocedural
  The difference in one of the complications of IHHT sessions (percent)
Fraction of inspired oxygen (FiO2) required for reducing cerebral tissue oxygenation based on near-infrared spectroscopy by 20% from the baseline (percent) | Periprocedural
  FiO2 is assessed in percent
Serum HIF-1α - hypoxia-inducible factor 1-alpha (pg/mL) | Baseline, Day 3, Day 4
  Serum HIF-1α is assessed in pg/mL
Serum NF-κB - nuclear factor-kappa B (ng/mL) | Baseline, Day 3, Day 4
  Serum NF-κB is assessed in ng/mL
Serum Nrf2 - Nuclear erythroid-related factor 2 (ng/mL) | Baseline, Day 3, Day 4
  Serum Nrf2 is assessed in ng/mL
HIF-1α - hypoxia-inducible factor 1-alpha in venous blood mononuclear cell nuclei (pg/mL) | Baseline, Day 4
  HIF-1α in venous blood mononuclear cell nuclei is assessed in pg/mL
NF-κB - nuclear factor-kappa B in venous blood mononuclear cell nuclei (ng/mL) | Baseline, Day 4
  NF-κB in venous blood mononuclear cell nuclei is assessed in ng/mL
Nrf2 - Nuclear erythroid-related factor 2 in venous blood mononuclear cell nuclei (ng/mL) | Baseline, Day 4
  Nrf2 in venous blood mononuclear cell nuclei is assessed in ng/mL
BIS ( Bispectral Index) monitoring (Units) | 6, 9, 15, 18, 24, 27, 33, 36, and 45 minutes from the initiation of the IHHT session
  The difference in BIS during IHHT sessions BIS is assessed in Units
PSV - Maximum peak systolic velocity measured by transcranial Doppler Ultrasound (cm/s) | Baseline, Day 4
  PSV is assessed in cm/s
Maximum peak T velocity measured by transcranial Doppler ultrasound (cm/s) | Baseline, Day 4
  peak T velocity is assessed in cm/s
TAMAX - time-averaged maximum velocity measured by transcranial Doppler ultrasound (cm/s) | Baseline, Day 4
  TAMAX is assessed in cm/s
TAMEAN - time-averaged mean velocity measured by transcranial Doppler ultrasound (cm/s) | Baseline, Day 4
  TAMEAN is assessed in cm/s
VF - volume flow measured by transcranial Doppler ultrasound (mL/s) | Baseline, Day 4
  VF is assessed in mL/s
RI - resistivity index measured by transcranial Doppler ultrasound (units) | Baseline, Day 4
  RI is assessed in Units
Peak velocity in the basal vein of Rosenthal on transcranial Doppler ultrasound (cm/s) | Baseline, Day 4
  Peak velocity is assessed in cm/s
PSV - peak systolic velocity in the middle cerebral artery (MCA) measured by transcranial Doppler ultrasound (cm/s) | Baseline, Day 4
  PSV is assessed in cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay O. Kamenshchikov, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.

REFERENCES:
- [Result] Uzun AB, Iliescu MG, Stanciu LE, Ionescu EV, Ungur RA, Ciortea VM, Irsay L, Motoasca I, Popescu MN, Popa FL, Pazara L, Tofolean DE. Effectiveness of Intermittent Hypoxia-Hyperoxia Therapy in Different Pathologies with Possible Metabolic Implications. Metabolites. 2023 Jan 25;13(2):181. doi: 10.3390/metabo13020181. PMID 36837800